CLINICAL TRIAL: NCT07349524
Title: Evaluation of the Efficacy and Safety of RSS0343 Tablets in Patients With Chronic Obstructive Pulmonary Disease (COPD): A Phase II, Randomized, Double-blind, Placebo-controlled Clinical Study.
Brief Title: A Study to Evaluate the Efficacy and Safety of RSS0343 Tablets in Patients With Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSS0343-202
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSS0343 tablets (Experimental)
  Interventions: Drug: RSS0343 tablets
- RSS0343 tablets Placebo (Placebo Comparator)
  Interventions: Drug: RSS0343 tablets Placebo

INTERVENTIONS:
Drug: RSS0343 tablets — RSS0343 tablets
  Arms: RSS0343 tablets
Drug: RSS0343 tablets Placebo — RSS0343 tablets Placebo
  Arms: RSS0343 tablets Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase II clinical trial designed to evaluate the efficacy and safety of RSS0343 tablets in patients with COPD. The study includes 3 study periods: a 4-week screening period, a 48-week treatment period, and a 4-week follow-up period. The primary endpoint is the annualized rate of moderate or severe exacerbations of COPD during the 48-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form.
2. Aged 40 to 80 years, male or female.
3. Body mass index (BMI) ≥18 kg/m².
4. Diagnosed with chronic obstructive pulmonary disease (COPD) as defined by the Chinese Guidelines for the Diagnosis and Management of COPD (2021 Revised Edition), with a documented COPD history of ≥12 months prior to screening.
5. Post-bronchodilator FEV₁/FVC <0.7 at the screening period; and post-bronchodilator FEV₁/FVC <0.7 with FEV₁% predicted ≥20% at baseline.
6. Documented history of at least ≥1 moderate or severe acute exacerbation of COPD (AECOPD) within 12 months prior to screening.
7. On stable doses of triple therapy or dual therapy for COPD maintenance treatment for ≥3 months prior to screening.
8. COPD Assessment Test (CAT) score ≥10 at randomization.
9. Current or former smoking history of ≥10 pack-years at screening.
10. Male and female subjects of childbearing potential and their partners must have no plans for conception or sperm/ova donation for 6 months (female subjects) or 3 months (male subjects) after the last dose and must voluntarily use effective contraception. Female subjects of childbearing potential must have a negative pregnancy test during screening and prior to the first dose and must not be lactating.

Exclusion Criteria:

1. Subjects with systemic immunosuppressants, biologic agents, or Th2 cytokine inhibitors within 12 weeks prior to randomization or within 5 half-lives of the drug, whichever is longer.
2. Subjects with medications known to potentially cause skin hyperkeratosis within 4 weeks prior to screening.
3. Subjects with the followings within 4 weeks prior to randomization: systemic corticosteroids, phosphodiesterase inhibitors, xanthine derivatives, leukotriene receptor antagonists, bacterial lysates, antitussive/expectorant medications, infusion of blood products or immunoglobulins.
4. Subjects with strong CYP3A inducers or inhibitors within 14 days or 5 half-lives (whichever is longer) prior to randomization.
5. Administration of live, attenuated live, or viral vector vaccines within 4 weeks prior to randomization.
6. Participation in another clinical trial involving an investigational product with active ingredients within 3 months prior to screening, or still within 5 half-lives of the investigational product at screening.
7. Prior treatment with RSS0343 tablets or treatment with products targeting the same mechanism of action within 3 months prior to screening.
8. History of lobectomy; or lung volume reduction surgery within 1 year prior to screening; or interventional procedures for chronic bronchitis within 1 year prior to screening.
9. Requirement for supplemental oxygen therapy for ≥15 hours per day or mechanical ventilation; or clinically significant sleep apnea requiring the use of a continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device.
10. Presence of a moderate or severe acute exacerbation of COPD (AECOPD) from 4 weeks prior to screening up to randomization.
11. Coexisting other respiratory or respiratory-related diseases.
12. Occurrence of pulmonary or other infections requiring systemic anti-infective therapy from 4 weeks prior to screening up to randomization.
13. Presence of autoimmune diseases mediated by eosinophils at screening.
14. Diagnosis of hypothyroidism, myxedema, chronic lymphedema, acromegaly, or livedo reticularis.
15. Diagnosis of psoriasis or lichen planus; Reiter's disease/keratoderma blennorrhagicum, keratoderma hemorrhagicum, or reactive arthritis; systemic lupus erythematosus, atopic dermatitis, chronic hand dermatitis, chronic contact dermatitis, or chronic psoriasis; chloracne, extensive verruca vulgaris, or keratotic dermatitis.
16. Known other severe medical conditions.
17. Laboratory tests, electrocardiogram (ECG), or other auxiliary examinations during the screening or baseline periods meeting the protocol-defined exclusion criteria.
18. Suspected or known hypersensitivity to the investigational product or any of its excipients.
19. Blood donation or blood loss ≥200 mL within 1 month prior to randomization, or ≥400 mL within 3 months prior to the first dose; or receipt of a blood transfusion within 8 weeks prior to the first dose; or difficulty with venipuncture, or physical condition unsuitable for intensive blood sampling.
20. Female subjects who are lactating, have a positive pregnancy test result, or plan to become pregnant during the study period.
21. History of drug abuse or substance abuse within 1 year prior to screening.
22. Any other medical or social reason deemed by the investigator to make the subject unsuitable for participation in the trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate or severe exacerbations of COPD during the 48-week treatment period | during the 48-week treatment period

SECONDARY OUTCOMES:
The annualized rate of moderate or severe exacerbations of COPD at week 12, 24, 36, and 48; | at week 12, 24, 36, and 48;
The time to first moderate or severe exacerbations of COPD at week 24 and 48; | at week 24 and 48;
The proportion of patients experiencing moderate or severe exacerbations of COPD at week 24 and 48 | at week 24 and 48
The change from baseline in pre- and post-bronchodilator forced expiratory volume in 1 second (FEV₁) at week 4, 8, 12, 24, 36, 48, and 52 | at week 4, 8, 12, 24, 36, 48, and 52
The change from baseline in pre- and post-bronchodilator forced expiratory volume in FEV₁% predicted at week 4, 8, 12, 24, 36, 48, and 52 | at week 4, 8, 12, 24, 36, 48, and 52
The change from baseline in pre- and post-bronchodilator forced expiratory volume in forced vital capacity (FVC) at week 4, 8, 12, 24, 36, 48, and 52; | at week 4, 8, 12, 24, 36, 48, and 52;
The change from baseline in the COPD Assessment Test (CAT) score at week 4, 8, 12, 24, 36, 48, and 52 | at week 4, 8, 12, 24, 36, 48, and 52
The change from baseline in the Evaluating Respiratory Symptoms in COPD (E-RS:COPD) score at week 4, 8, 12, 24, 36, 48, and 52 | at week 4, 8, 12, 24, 36, 48, and 52
The change from baseline in the St. George's Respiratory Questionnaire (SGRQ) score at week 4, 8, 12, 24, 36, 48, and 52; | at week 4, 8, 12, 24, 36, 48, and 52;
The proportion of patients with a SGRQ response (a ≥4-point decrease from baseline) at week 48; | at week 48;

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided